CLINICAL TRIAL: NCT01572077
Title: Rt Ventricular Substrate Metabolism as a Predictor of Rt Heart Failure in Patients With Pulmonary Arterial Hypertension
Acronym: RVMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Lisa Mielniczuk, Co- Medical Director Pulmonary Hypertension Clinic, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2010539-01H
Record Dates: First submitted 2012-03-29; First posted 2012-04-05 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — 14-fluoro-6-thiaheptadecanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FTHA/GDF PET imaging (Experimental): This study plans to enrol 60 subjects with Type I pulmonary arterial hypertension (PAH) and 20 healthy, age and sex individuals to serve as normal controls. These subjects will have no known cardiac or pulmonary disease.
  Both groups will undergo FTHA/FDG PET imaging.
  Interventions: Radiation: FTHA, FDG PET imaging.

INTERVENTIONS:
Radiation: FTHA, FDG PET imaging. — Subjects will undergo PET scans on 2 different days using 2 separate tracers, FTHA(fluoro-6-this-hepadecanoic acid) and FDG(fluoro-2- deoxy-glucose).

SUMMARY:
The purpose of this study is to evaluate patterns of metabolic activity in the heart of patients with pulmonary arterial hypertension(PAH). Patients with PAH are at risk of developing weakness or failure of the right side of the heart.It is possible that there is a relationship between the development of heart failure and the way the heart uses energy sources, such as sugar. This study is designed to evaluate the way the heart uses sugar uptake in patients with PAH using positron emission tomography(PET imaging)

DETAILED DESCRIPTION:
PAH results in premature death as a result of right ventricular dysfunction. However, there are substantial differences among patients in their tendency to develop right heart failure. This study proposes to determine if right ventricular (RV) changes can predict the development of right heart failure in patients with PAH.

In addition, the study aims to evaluate the relationship of right ventricular metabolism to other physiologic responses in PAH,including:pulmonary vascular resistance, serum BNP and changes in cardiac hypertrophy and function. In conjunction with hemodynamic measurements, biomarkers and cardiac magnetic resonance imaging (MRI); RV metabolism will be evaluated with (18F) FTHA and (18F)FDG cardiac PET imaging.

A cohort of 20 age sex matched individuals will serve as normal controls. These subjects will have no known cardiac or pulmonary disease with normal ventricular function and estimates pulmonary pressures on echocardiogram.

ELIGIBILITY:
Inclusion Criteria:(PATIENTS)

* Patients with diagnosis of Category 1 pulmonary arterial hypertension due to any of the following: idiopathic, familial, associated with connective tissue disease, HIV disease or anorexigen use.
* All patients who will require a right heart catheterization for further clinical management and/or diagnosis.
* Patients will be considered eligible if they have no significant coronary artery disease (stenosis > 70% in a proximal or mid major coronary artery) or moderate coronary artery disease (60-70%) with abnormal left ventricular function (EF<50%)
* Patients will be considered eligible in the absence of current or recent evidence of right heart failure.
* No previous hospital admission or requirements of intravenous diuretics for right heart failure within 6 months of enrolment.
* No increase in oral diuretics to control fluid volume within 6 months prior to enrolment
* No current symptoms and signs of fluid retention or right heart strain, including any of the following: development of new ascites or peripheral edema > = 2+, JVP >7 cm above the sternal angle or a right atrial pressure >14 mmHg at the time of right heart catheterization.
* In addition, we will include a small cohort of up to 15 patients with PAH and current RHF.

Exclusion Criteria:

* Patients with known significant coronary artery disease(defined as known stenosis >70% in a proximal or mid major artery or moderate coronary artery disease (60-70%)in a coronary artery and associated left ventricular ejection fraction <50%.
* Patients with diabetes mellitus who require the use of oral hypoglycemics and or insulin.
* Implantable metal devices, incompatible with magnetic resonance imaging.
* Other contraindications of magnetic resonance imaging.

Normal Control Subjects:

* Subjects will have no known cardiac or pulmonary disease.
* Normal ventricular function and estimated pulmonary pressures on echocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary death OR clinical right heart failure hospitalization | 1year
  Clinical RHF admission requiring ONE of the following:intravenous diuretics or an increase in oral diuretics >50%of baseline for at least 7 days.

SECONDARY OUTCOMES:
Change in right ventricular size and function as measured by cardiac MRI, between baseline and 1 year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Mielniczuk, MD, Principal Investigator — University of Ottawa Heart Institiute
Locations (1):
- University of OttawaHeart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided